CLINICAL TRIAL: NCT05612971
Title: iAmHealthy Parents First: A Televideo Parent and Child Obesity Program for Rural Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00147611; R01NR019810 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Weight Loss; Pediatric Obesity
MeSH Terms: conditions — Weight Loss; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iAmHealthy Parents First (Experimental): iAmHealthy Parents First families will take part in a group program with other adults over Zoom. Children will not be involved during this time. Adults will participate in these group sessions weekly for three months. Each meeting will last approximately an hour. Fifteen dyads from each cohort will be randomized to the iAmHealthy Parents First group.
  After 3 months, both iAmHealthy Parents First and iAmHealthy families will take part in an educational group program with parents and their children. These meetings will be focused on living healthy lifestyles and engaging in healthy habits as a family and will occur three weeks out of four for four months. There will be three additional family-based group sessions spread over the final two months of the program. iAmHealthy Parents First adults will continue to meet monthly during the family-based program (on weeks when the family-based group does not meet) to continue the adult program.
  Interventions: Behavioral: iAmHealthy Parents First
- iAmHealthy (Active Comparator): iAmHealthy families will receive an informational newsletter once a month for three months. This group will be given the flexibility to start their weight loss journey using self-guided methods. No formal group sessions will be provided for three months. Fifteen dyads from each cohort will be randomized to the iAmHealthy group.
  After 3 months, both iAmHealthy Parents First and iAmHealthy families will take part in an educational group program with parents and their children. These meetings will be focused on living healthy lifestyles and engaging in healthy habits as a family and will occur three weeks out of four for four months. There will be three additional family-based group sessions spread over the final two months of the program.
  Interventions: Behavioral: iAmHealthy

INTERVENTIONS:
Behavioral: iAmHealthy Parents First — iAmHealthy Parents first is a 3-month adult obesity treatment program targeting the unique needs of adults with school-age children. Following the iAmHealthy Parents First program, these dyads will take part in a 6-month family-based healthy lifestyles program.
  Arms: iAmHealthy Parents First
Behavioral: iAmHealthy — The iAmHealthy group will receive newsletters for three months. Following this period, these dyads will take part in a 6-month family-based healthy lifestyles program.
  Arms: iAmHealthy

SUMMARY:
The purpose of this study is to assess whether providing a parent-only group program before providing a parent and child group program works better than the parent and child group program alone.

DETAILED DESCRIPTION:
The goal of this project is to determine if an adult intervention followed by a family-based program (iAmHealthy Parents First) will result in a larger percentage of weight loss in parents and children compared to solely a family-based program (iAmHealthy). Furthermore, the investigators aim to discover if administering iAmHealthy Parents First will improve dietary intake, physical activity, and weight-related quality of life among parents and children when compared to iAmHealthy. Parent/child dyads will be recruited from rural elementary schools, medical clinics, and organizations across Kansas and neighboring states.

ELIGIBILITY:
Inclusion Criteria:

* Family lives in a rural area (city and/or county population <20,000) or as defined by RUCA codes, Urban Influence Codes, amount of agricultural income, or individual commuting patterns
* Child BMI%ile ≥ 85th and parent BMI 25-50 kg/m2
* Child in 1st-5th grade or 6-11 years of age
* Child and parent speak English
* Family is available at times intervention is offered

Exclusion Criteria:

* For parents: new MI, stroke or cancer diagnosis in past 6 months, recent bariatrics surgery (within 2 years) or planned within 1 year, pregnancy in last 6 months or planned within 1 year

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent weight change in parents and BMIz (BMI z-score) in children | Baseline, 3 months, 9 months
  Parents and children will measure body weight on a study-provided digital scale following instructions provided by study team.

SECONDARY OUTCOMES:
Mediator: Attendance | Baseline, 3 months, 9 months
  Group and individual session attendance (percent of sessions) will be tracked on REDCap, a secure, web-based application designed exclusively to support data capture for research studies.
Mediator: Reciprocal modeling | Baseline, 3 months, 9 months
  Reciprocal influence (parent response as mediator for child; child response as mediator for parent) will be operationalized as adult or child weight loss.
Moderator: Family functioning | Baseline, 3 months, 9 months
  Family functioning will be measured using the Family Assessment Device (FAD). This is the gold-standard measure of structural, organizational, and transactional characteristics of families including general family functioning (core scale of interest) and 6 additional subscales: affective involvement, affective responsiveness, behavioral control, communication, problem solving, and roles. This questionnaire will be completed by adults. The FAD is scored by adding responses of each scale (1 - 4) and dividing by the number of items in each scale (between 6 - 12). The higher the overall score, the worse the level of family function.
Moderators: Genetic casual attributions | Baseline, 3 months, 9 months
  Genetic casual attributions will be measured using a a 2-item Likert scale that assesses perceived genetic role for weight status and potential for weight loss. This will be completed by adults. Those who endorse completely or mostly for the role of genes in weight loss will be characterized as having "high genetic attribution" for weight status.

OTHER OUTCOMES:
Participation rates and representativeness of school and clinic samples | 9 months
  Reach (participation rates and representativeness) will be assessed at primary care versus school settings. Participation rates will be calculated in multiple ways to include: 1) the percentage of individuals on lists who respond and 2) the percentage of eligible respondents who enroll. Enrolled participants will be classified as recruited from the school or clinic according to participant self-report of how they heard about the study, or if recruited from both channels, which one had the most influence on their participation. Representativeness will be assessed by comparing demographics (age/grade, sex, race/ethnicity, BMI where available) between enrolled participants and non-participants including 1) potential participants on recruitment lists and 2) those who are screened but do not enroll. In addition, the investigators will assess the impact of nurse engagement/leadership on participant reach and attendance.
The impact of nurse engagement/leadership on participant reach and attendance as measured by the Community Engagement Survey and semi-structured interviews | 1 month and 10 months
  The Community Engagement Survey will assess nurse engagement and leadership, which is divided into seven separately summed subscales. Interview data collection and analysis will be led by Co-I who has the necessary training/experience to conduct semi-structured interviews, with assistance from members of the research team. Dedoose will be used to assist the researchers in efficient and organized data storage, coding, retrieval, comparing, and linking.
Physical activity | Baseline, 13 weeks, 14 weeks, 15 weeks, 16 weeks/4 months, 18 weeks/5 months, 6 months, 7 months, 8 months, 9 months
  This measure will be completed on a subset of participants. The Garmin activity device is a consumer wearable that will automatically detect and track activity such as walking, running, and cycling. This device will measures steps. Self-reported physical activity will be collected from the exercise vital sign.
Child diet | Baseline, 13 weeks, 14 weeks, 15 weeks, 16 weeks/4 months, 18 weeks/5 months, 6 months, 7 months, 8 months, 9 months
  This measure will be completed on a subset of participants. Child diet will be parent reported using the Children's Eating Habits Questionnaire-Food Frequency Questionnaire section (CEHQ-FFQ). We are interested in the frequency of red foods ("junk" foods) and fruits/vegetables.
Child pain | Baseline, 13 weeks, 14 weeks, 15 weeks, 16 weeks/4 months, 18 weeks/5 months, 6 months, 7 months, 8 months, 9 months
  This measure will be completed on a subset of participants. Child pain will be measured using the Pediatric Pain-Short form questionnaire from the Patient Reported Outcomes Measurement information system (PROMIS). Scores are summed and converted to T-scores using a conversion table. A T-score of 50 with a standard deviation of 10 is considered the mean. A minimally important difference in T-score is 3 points.
Home environment | Baseline, 13 weeks, 14 weeks, 15 weeks, 16 weeks/4 months, 18 weeks/5 months, 6 months, 7 months, 8 months, 9 months
  This measure will be completed on a subset of participants. Home environment will be assessed through the Confusion, Hubbub, and Order Scale (CHAOS). Applicability of statements to respondent's own home environment is rated on a 4-point Likert-type scale: 1 (not at all), 2 (a little bit), 3 (somewhat), or 4 (very much). The range of scores is 15-60 with higher scores indicating a more negative home environment. Previous studies have grouped CHAOS scores into categories (low: <25; moderate/low: 25-30; moderate/high: 31-35; high: >35).
Caregiver stress | Baseline, 13 weeks, 14 weeks, 15 weeks, 16 weeks/4 months, 18 weeks/5 months, 6 months, 7 months, 8 months, 9 months
  This measure will be completed on a subset of participants. Caregiver stress will be assessed using the Perceived Stress Scale. Data will be analyzed/interpreted as a continuous variable and a categorical value. Responses to the scale are reported as a continuous variable (scores ranging from 0-47) and can be interpreted into one of three levels: low stress (scores 0-13), moderate stress (scores 14-26), or high stress (scores 27- 40). Higher scores correspond to higher levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Davis, PhD, MPH, Principal Investigator — University of Kansas Medical Center; Christie Befort, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Davis AM, Befort CA, Lancaster BD, Tuck C, Polivka BJ, Carlson JA, Fleming K, Romine RS, Dean K, Murray M. Rationale and design of integrating a parents first obesity intervention with a pediatric weight management intervention for rural families - Evaluating the ripple effect. Contemp Clin Trials. 2023 May;128:107140. doi: 10.1016/j.cct.2023.107140. Epub 2023 Mar 7. PMID 36893988
- See also: Study website — http://www.iamhealthyparentsfirst.org